CLINICAL TRIAL: NCT01742884
Title: Evaluation of the Efficacy and Safety of a Treatment for Dry Eye Syndrome: Thealoz
Brief Title: Efficacy and Safety of a Treatment for Dry Eye Syndrome: Thealoz
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto Universitario de Oftalmobiología Aplicada (Institute of Applied Ophthalmobiology) - IOBA (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IOBA-Thea-001-2012
Record Dates: First submitted 2012-12-04; First posted 2012-12-06 (Estimated); Last update posted 2015-01-08 (Estimated); Status verified 2015-01

CONDITIONS: Moderate Dry Eye Syndrome
Keywords: Dry Eye Syndrome
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Trehalose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Thealoz (Experimental): Treatment with Thealoz (Trehalose) 3% for 1 month
  Interventions: Other: Thealoz
- Treatment with Thealoz´s vehicle (Placebo Comparator): Treatment with Thealoz´s vehicle for 1 month
  Interventions: Other: Vehicle

INTERVENTIONS:
Other: Thealoz — Instillation of 1 drop of Thealoz
  Other Names: Thealoz, Trehalose
  Arms: Thealoz
Other: Vehicle — 1 drop of the vehicle will be instillated in the eye
  Other Names: Instillation of Thealoz´s vehicle
  Arms: Treatment with Thealoz´s vehicle

SUMMARY:
The purpose of this study is to determine if Thealoz is effective in Dry Eye Syndrome exposed to controlled adverse environmental conditions.

ELIGIBILITY:
Inclusion Criteria:

* Man/woman ≥ 18 years old, able to freely give consent to participate in the study
* Fluorescein corneal staining ≥ 1 and ≤ 3 in Oxford Scales
* At least 2 of the following tests altered:
* Ocular Surface Disease Index (OSDI) Test symptoms between 12 and 40
* BUT ≤10 seconds
* Lissamine green conjunctival staining ≥ 1
* Schirmer Test without anesthesia ≤ 5 mm
* Informed consent signed
* Data protection consent signed

Exclusion Criteria:

* Sensitivity or known intolerance to any of the product used in the study
* Story of ocular infections or severe ocular inflammation within the 6 previous months to study inclusion
* Any active ocular pathology other than Dry Eye Syndrome
* Any traumatize or ocular surgery that may affect corneal sensitivity and/or normal tear distribution (e.g. cataract surgery, refractive surgery) within the 6 previous months to study inclusion
* Use of contact lenses in the 3 previous months to study inclusion
* Use of any ocular topical medications other than the treatment for Dry Eye Syndrome
* Ocular treatment for Dry Eye Syndrome with corticosteroids 1 month before inclusion visit or Cyclosporin A 3 months before inclusion
* Diagnosis of Rosacea or Severe Blepharitis (associated to systemic or ocular pathologies) Any severe uncontrolled systemic disease that may affect the eye (except for primary or secondary Sjögren)
* Start, discontinuation or change within the study of the dosage of antihistaminics, cholinergic agents, beta blockers, anti depressants or any other systemic drugs with potential effects in the tear film
* No pregnant or breastfeeding women is allowed to participate in the study. Childbearing potential women must use contraceptive means during the whole study.
* Participation in another clinical trial in the last 30 days before study inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-12; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with fluorescein corneal staining reduction of at least 1 point | 1 Month
  Proportion of subjects with staining reduction within the treatment group vs proportion of staining reduction in control group

SECONDARY OUTCOMES:
Best Corrected Visual Acuity | 1 month
  Best Corrected Visual Acuity at Exit visit compared to baseline visit
Intraocular pressure | 1 month
  Pathological elevations of intraocular pressure from baseline
Eye fundus alterations | 1 month
  Presence of any pathological finding in eye fundus while the patient is in the study
Corneal Pachymetry | 1 month
  Changes in corneal thickness along the study

CONTACTS AND LOCATIONS:
Overall Officials: Maria Jesus Gonzalez, PhD, Principal Investigator — IOBA - University of Valladolid
Locations (1):
- IOBA - University of Valladolid, Valladolid, Valladolid, Spain